CLINICAL TRIAL: NCT01237574
Title: Multicentre Prospective Cohort Study of Patients With Chronic Alcoholic and/or Metabolic Liver Disease
Acronym: CALMET
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2010/38
Record Dates: First submitted 2010-10-25; First posted 2010-11-09 (Estimated); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Liver Diseases, Alcoholic; Metabolic Diseases
Keywords: Liver Diseases; Alcoholic; Metabolic Diseases; cohort; liver disease
MeSH Terms: conditions — Liver Diseases, Alcoholic; Metabolic Diseases; Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * serum
  * plasma (DNA)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: Patients with chronic alcoholic and/or metabolic liver disease
  Interventions: Other: Intervention according to the standard of care.

INTERVENTIONS:
Other: Intervention according to the standard of care. — Every 6 months, patients will have clinical, biological and morphological evaluation according to the standard of care.

SUMMARY:
Chronic alcoholic and metabolic liver diseases are the two main liver diseases in France. The long-term prognosis of these two diseases are not well known because main studies are retrospective and with only alcoholic patients. The knowledge of the natural history of these diseases should improve the management of patients with such diseases.

The aim of this prospective cohort is to describe the natural history of patients with chronic liver disease due to alcohol or metabolic disease and to identify factors associated with complications of these liver diseases (cirrhosis, hepatocellular carcinoma, ascites. ..).

DETAILED DESCRIPTION:
In 2010, the two most frequent chronic liver diseases are alcoholic and metabolic disease. The natural history of these two diseases is not well known. Indeed, most of the studies were retrospective and evaluated alcoholic disease or metabolic disease but never both diseases. However, these two diseases have the same histological lesions and can be associated. The knowledge of the natural history of these diseases could improve the management of patients in order to decrease complications and improve survival. The aim of this prospective study is to describe the natural history of chronic liver disease due to alcohol and/or metabolic syndrome and to identify factors associated with complications (ascites, encephalopathy, death, complications of obesity, diabetes or chronic alcohol abuse). All patients will be followed every 6 months for 3 years with clinical, biological and morphological parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* chronic liver disease (liver biopsy with bridging fibrosis or cirrhosis) or non-invasive markers of fibrosis (fibrotest > 0.58, FibroScan > 7.9 kPa)
* no decompensated cirrhosis
* chronic alcohol use and/or metabolic syndrome (at least 3 criteria of metabolic syndrome)
* Written informed consent
* Patient covered by the French health insurance system

Exclusion Criteria:

* short term life threatening disease
* Other cirrhosis causes
* Impossibility of regular follow-up
* Under guardianship major Patient
* Presence of focal hurt suggestive of CHC
* pregnant women
* cirrhosis complication
* Child-pugh score superior or equal to 7

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years old patient with chronic liver disease (liver biopsy with bridging fibrosis or cirrhosis) or non-invasive markers of fibrosis (fibrotest > 0.58, FibroScan > 7.9 kPa), no decompensated cirrhosis, chronic alcohol use and/or metabolic syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2010-11-23 (Actual); Primary Completion 2020-12-12 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Death | up to 84 months

SECONDARY OUTCOMES:
Complications of liver disease | up to 84 months
  ascites, encephalopathy, liver cancer, bleeding from oesophageal varices
Complications of obesity | up to 84 months
  cardiovascular diseases, pulmonary diseases, etc.
Complications of diabetes | up to 84 months
  renal failure,etc.

CONTACTS AND LOCATIONS:
Locations (36):
- France (36):
  - CHU d'Angers, Angers
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - CH Pierre Oudot, Bourgoin
  - CHU de Brest - Hôpital La Cavale Blanche, Brest
  - CHU de Caen, Caen
  - CH de Chateauroux, Châteauroux
  - CHU Clermont-Ferrand - Hôpital Estaing, Clermont-Ferrand
  - CH Laennec, Creil
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble
  - CH Le Mans, Le Mans
  - GH-ICL - Hôpital Saint Philibert, Lille
  - CH de Limoges - Hôpital Dupuytren, Limoges
  - HCL - Hôpital Hôtel Dieu, Lyon
  - APHM - Hôpital La Conception, Marseille
  - Hôpital Saint-Joseph, Marseille
  - CH de Montauban, Montauban
  - CHU de Nancy - Hôpital de Brabois, Nancy
  - CHU de Nice - Hôpital Archet 2, Nice
  - Hôpital Carémeau, Nîmes
  - CHR Orléans - Hôpital La Source, Orléans
  - APHP - Hôpital Bicêtre, Paris
  - APHP - Hôpital Jean Verdier, Paris
  - APHP - Hôpital Paul Brousse, Paris
  - APHP - Hôpital Pitié Salpetrière, Paris
  - APHP - Hôpital Saint-Antoine, Paris
  - APHP - Hôpital Tenon, Paris
  - APHP Hôpital Cochin, Paris
  - APHP- CHU Henri Mondor, Paris
  - CH de Perpignan - Hôpital Saint-Jean, Perpignan
  - CHU de Bordeaux - Hôpital du Haut-Lévêque, Pessac
  - CHRU de Poitiers, Poitiers
  - CHU de Reims - Hôpital Robert Debré, Reims
  - CHU de Rouen, Rouen
  - CHRU de Strasbourg - Nouvel Hôpital Civil, Strasbourg
  - CHU de Toulouse - Hôpital Purpan, Toulouse
  - CHRU de Tours - Hôpital Trousseau, Tours